CLINICAL TRIAL: NCT00271193
Title: A Primary Care Intervention for Weight Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT00271193; K24DK065018 (NIH); NCT00271193 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2005-12-29; First posted 2005-12-30 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Healthy

ARMS (2):
- 1 (No Intervention): Control group, receives physician advice for weight loss and materials
- 2 (Active Comparator): Active treatment group, receives physician advice, materials, and brief weight loss counseling
  Interventions: Behavioral: Weight loss counseling

INTERVENTIONS:
Behavioral: Weight loss counseling — A comparison of weight loss advice provided by primary care physicians to advice plus brief weight loss counseling provided by medical assistants. Participants in both groups receive weight loss materials.
  Arms: 2

SUMMARY:
The study will test whether adding brief counseling visits with an ancillary health care provider (a nurse or nursing assistant) will induce additional weight loss, as compared with quarterly physician visits alone. All visits will take place at the site of usual patient care (i.e., the primary care clinic).

ELIGIBILITY:
Inclusion Criteria:

Body mass index (BMI) of 27 to 50 kg/m2 Capacity to provide informed consent Ability to find transportation to and from counseling sessions Willingness to be randomized to either program Commitment to attend all sessions and to complete study-related assessments, including blood tests and questionnaires

Exclusion Criteria:

Type I diabetes Myocardial infarction or stroke within the previous 6 months Clinically significant renal or hepatic disease (as judged by a study physician) History of cancer in the past 5 years Congestive heart failure requiring diuretics Previous weight loss surgery Endocrine conditions that may cause weight gain, including unstable thyroid disease or hypercortisolism Initiation of therapy with or dose change to any of the following medications within 6 weeks of starting the study: insulin; metformin; sulfonylurea; thiazolidinedione; HMG-CoA reductase inhibitor ("statin"); or SSRI for depression Long-term use of any of the following medications: oral or high-dose inhaled steroid; atypical antipsychotic; tricyclic antidepressant; antiepileptic; any prescription or over-the-counter drug for weight loss Systolic blood pressure > 160 or diastolic blood pressure > 100 Hemoglobin A1c ≥ 10 Pregnancy or lactation Clinically significant psychiatric disease, including major depression, eating disorders, or substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Weight change | 6 months

SECONDARY OUTCOMES:
Blood pressure | 6, and 12 months
Lipids | 6, and 12 months
Fasting glucose | 6, and 12 months
Quality of life | 6, and 12 months
Weight change | 12 months
Waist circumference | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Wadden, PhD, Principal Investigator — Director, Weight and Eating Disorders Program, University of Pennsylvania
Locations (2):
- United States (2):
  - Edward S. Cooper Internal Medicine Practice, Philadelphia, Pennsylvania
  - Presbyterian Medical Group, Philadelphia, Pennsylvania